CLINICAL TRIAL: NCT01097408
Title: A Randomised, Double-Blind, Placebo-Controlled Study to Determine the Pharmacokinetics, Safety and Tolerability of AZD7295 Capsules in Healthy Volunteers
Brief Title: Pharmacokinetics of AZD7295 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrow Therapeutics (Industry)
Responsible Party: Liz Clark, Arrow Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCV689-105
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD7295 (Experimental)
  Interventions: Drug: AZD7295
- Matched placebo (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: AZD7295 — Up to 650mg AZD7295 capsules per dose. To be given 2 or 3 times daily for 5 days.
  Arms: AZD7295
Drug: Placebo comparator — Placebo capsules
  Arms: Matched placebo

SUMMARY:
This is a pharmacokinetics (PK) and safety study of AZD7295 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers, aged 18-65 years.

Exclusion Criteria:

* Previous exposure to AZD7295, clinically relevant disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of AZD7295 capsules | 0-72h after each dose
  PK parameters of AZD7295 will be measured after single and repeated doses (AUC, Cmax, t1/2)

SECONDARY OUTCOMES:
Safety and tolerability of AZD7295 capsules | 0-72h after each dose
  Safety and tolerability of AZD7295 will be assessed after single and repeated doses (adverse events, ECGs, vital signs, safety laboratory tests)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Collier, Mb ChB, Principal Investigator — Quotient Clinical Research
Locations (1):
- Quotient Clinical Research, Nottingham, United Kingdom